CLINICAL TRIAL: NCT06486389
Title: The Effect of Reading Fairy Tales and Coloring on Children's Fear Level and Parental Health Care Satisfaction in Children Aged 3-6 Years Who Are Administered Inhaler Drugs
Brief Title: The Effect of Reading Fairy Tales and Coloring on Children's Fear Level in Children Who Are Administered Inhaler Medication With a Mask.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Nuray Macuncu, Nurse, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TÜTF-GOBAEK 2022/318
Record Dates: First submitted 2024-03-12; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Fear Anxiety; Satisfaction
Keywords: Inhaler medicine; Fear; Readin Fairy Tales; Coloring; Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Chromosome Painting

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: None (Open Label) Primary Purpose: Supportive Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- distraction methods (Experimental): reading fairy tales
  Interventions: Device: reading fairy tales
- distraction method (Experimental): painting
  Interventions: Device: painting
- Control Grup (No Intervention): Routine Treatment Group

INTERVENTIONS:
Device: reading fairy tales — Reading fairy tales during inhaler medication administration.
  Arms: distraction methods
Device: painting — painting during inhaler medication administration
  Arms: distraction method

SUMMARY:
This thesis study was conducted as an unblinded, randomized controlled experiment to examine the effects of reading and coloring fairy tales, which can be used during inhaler medication administration with a mask, on children's fear level and parental health care satisfaction.

DETAILED DESCRIPTION:
Data were collected at Edirne Sultan 1. Murat State Hospital Pediatrics Clinic between September 2023 and January 2024. Children aged 3-6 were included in the study. In the research, the sample was divided into three groups. 99 children participated in the study, 33 children in each group. Using the randomization program, it was determined which sample group the children would be included in.

In the study, reading fairy tales and coloring were used as distraction methods for the experimental group. Inhaler medication was administered via mask to the control group without any application. The implementation period of the research lasted an average of four months. Necessary ethical permissions were obtained before the research. In the study, the Child Fear Scale was used to measure the level of fear, the PedsQL Health Care Satisfaction Scale was used to measure parental satisfaction, and the Children's Emotional Indicators Scale was used to measure emotional indicators. Explanatory information about the application was given to the children and their parents by the researcher, and they were voluntarily informed and signed a consent form. Research data were collected by the researcher by meeting children and parents face to face.

ELIGIBILITY:
Inclusion Criteria:

1. Parent and child volunteering to participate in the study,
2. The child is between the ages of 3-6,
3. Being admitted due to respiratory system disease,
4. Inhaler treatment with a mask will be applied.

Exclusion Criteria:

1. Parent and child not voluntarily participating in the study,
2. The child has any genetic, congenital, chronic or metabolic disease,
3. The child has vision, hearing and speech problems,
4. The child's vital signs are unstable (no fever, tachypnea, etc.) and the need for any emergency intervention.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Personal data collection form | baseline
  The data collection form was prepared by the researchers in line with the literature. In this form 8 questions about the characteristics of children.There are 18 questions in total, 10 of which include parent and family characteristics.
Child Fear Scale | baseline
  The scale was developed to determine the anxiety level of children aged 5-10 years. There are various facial expressions in the scale and a numerical value is given for each facial expression. The lowest score obtained from the scale is "0" and the highest score is "4". The higher the score obtained from the scale, the higher the level of anxiety felt in the child. The inhaler was filled by the child before medication administration.
Child Emotional Manifestation Scale | baseline
  In the scale, emotional indicators are evaluated in terms of 5 parameters. These parameters are; facial expression, voice, activity, interaction and cooperation level. These five parameters are scored from 1 to 5, and the lowest "5" and the highest "25" points are obtained at the end of the evaluation of the scale. A low score from the scale indicates a positive emotional state, and an increase in a score indicates a negative emotional state. The inhaler was filled out by the researcher before drug administration.

SECONDARY OUTCOMES:
Child Fear Scale | within 10 minutes after inhaler treatment
  In the scale, emotional indicators are evaluated in terms of 5 parameters. These parameters are; facial expression, voice, activity, interaction and cooperation level. These five parameters are scored from 1 to 5, and the lowest "5" and the highest "25" points are obtained at the end of the evaluation of the scale. A low score from the scale indicates a positive emotional state, and an increase in a score indicates a negative emotional state. the inhaler was filled by the child within 10 minutes of treatment
Child Emotional Manifestation Scale | within 10 minutes after inhaler treatment
  In the scale, emotional indicators are evaluated in terms of 5 parameters. These parameters are; facial expression, voice, activity, interaction and cooperation level. These five parameters are scored from 1 to 5, and the lowest "5" and the highest "25" points are obtained at the end of the evaluation of the scale. A low score from the scale indicates a positive emotional state, and an increase in a score indicates a negative emotional state. inhaler was filled by the researcher within 10 minutes of treatment
PedsQL Health Care Parental Satisfaction Scale | within 10 minutes after inhaler treatment
  This scale was created to evaluate parents' satisfaction with health care and to increase the level of satisfaction with health care; It consists of six subheadings and 25 questions: information, family participation, communication, technical skills, emotional needs and general satisfaction. The statements in the PedsQL Health Care Satisfaction Scale are; never satisfied = 0, sometimes satisfied = 25, It was quantified with a score of most of the time = 50, almost always satisfied = 75, always satisfied = 100 points. inhaler filled by parent within 10 minutes of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- TÜRKİYE, Edirne, Merkez, Turkey (Türkiye)